CLINICAL TRIAL: NCT04160273
Title: Evaluation of Postpartum Posttraumatic Stress Disorder at Angers University Hospital (ESPT-PP)
Acronym: ESPT-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-A02369-48
Record Dates: First submitted 2019-11-05; First posted 2019-11-12 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Delivery; Post Partum
Keywords: Posttraumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnosis and follow-up arm (Experimental): Patients are informed during the 9th month pregnancy consultation at Angers University Hospital by the midwife or obstetrician in charge of the consultation. They are included in the 48 hours following the delivery after their hospitalization in the maternity ward.
  During hospitalization, socio-demographic and medical data are collected and the Peritraumatic Distress Inventory, the peritraumatic dissociation questionnaire and the Edinburgh peritraumatic dissociation questionnaire are completed before returning home.
  Follow-up at 1 month and 1 year is carried out by the investigators and the patient answers to the PCL-S questionnaire. Also collected during this call are information on the physical and mental state of the patient, the state of health of her newborn and the progress of the return home.
  Patients are considered at high risk of PTSD if they have a PCL-S score ≥ 26 at 1 month. A consultation with a psychiatrist is offered to these patients at risk of PTSD.
  Interventions: Diagnostic Test: patient questionnaire and telephone follow-up

INTERVENTIONS:
Diagnostic Test: patient questionnaire and telephone follow-up — PDI scale is filled in before returning home and follow-up at one month and one year thanks to a telephone call during which the patient answers the PCL-S questionnaire

SUMMARY:
The purpose of this study is to estimate the prevalence of post-traumatic stress disorder (PTSD) at one month in women who have given birth at the University Hospital of Angers over a period of 1 year.

DETAILED DESCRIPTION:
Childbirth is a natural process expected, prepared and imagined by all future parents.

A traumatic experience of childbirth and its consequences is a major problem that is often underestimated for women's health. Some women may develop Post Traumatic Stress Disorder (PTSD) after delivery. The literature reports a prevalence of PTSD in relation to childbirth of 1.3 to 6%.

Symptoms of post-traumatic stress can be triggered by any event, perceived as threatening to the life or physical integrity of the person or a third party and causing intense fear, helplessness and horror.

It may be thought that childbirth, by its psychological and physiological characteristics, can be described as an extreme experience and its experience depends on multiple factors. Thus, an innocent childbirth for caregivers can be traumatically experienced by the woman.

The symptoms described are symptoms of avoidance (inability to return to the scene of trauma, denial of trauma), symptoms of intrusion (nightmares, reviviscences) and symptoms of neuro-vegetative hyper activation (sleep disorders, anger, emotional indifference ).

The development of PTSD following childbirth is a known phenomenon, but minimized and very little diagnosed by obstetric teams.

Therefore, it seems interesting to assess the prevalence of PTSD during childbirth in order to optimize our management, that is to identify patients at risk of PTSD and offer them adapted psychological follow-up.

This study also aims to describe the kinetics of the development of post-traumatic postpartum symptoms and to study the risk factors for the development of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Major and francophone patient,
* Giving birth (≥ 37 weeks of amenorrhea) to the maternity hospital of Angers University Hospital,
* Agree to participate in the study (signature of consent).

Exclusion Criteria:

* Birth of a child born lifeless,
* Patient deprived of liberty by judicial or administrative decision,
* Patient subject to a legal protection measure,
* Patient unable to express her consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1451 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
The risk of PTSD at 1 month is detected using the PCL-S scale. | 1 Month
  The risk of PTSD at 1 month is detected using the PCL-S scale. Patients are considered at high risk if they have a score ≥ 26 on this scale. A consultation with a psychiatrist is offered to these patients at risk of PTSD in order to make the diagnosis and offer them appropriate care if necessary.

SECONDARY OUTCOMES:
Determine the emotional distress of a person at the time of a traumatic event at 1 month and one year | 1 month and 1year
  Using the immediate postpartum PDI scale at 1 month and one year
Detect a state of post-traumatic stress | 1 Month and 1 year
  Using the PCL-S scale at 1 month and 1 year
Collect the risk factors associated with PTSD | 5 Days
  The risk factors studied are as follows: socio-economic status, gestational-parity, obstetrical history, psycho-pathological antecedents, addictions , current pregnancy course, term childbirth, mode of delivery and its complications, course of the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEGENDRE, MDPhD, Principal Investigator — University Hospital, Angers
Locations (1):
- UH Angers, Angers, France